CLINICAL TRIAL: NCT03766178
Title: A Single-arm, Open Phase II Clinical Trial of Anti-PD-1 Antibody SHR-1210 Combined With Nimotuzumab as Second-line Treatment of Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Study of Anti-PD-1 Antibody SHR-1210 Plus Nimotuzumab in the Treatment of Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Director, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FQX-002
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — nimotuzumab; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab + SHR-1210 (Experimental): Nimotuzumab + SHR-1210
  Interventions: Drug: Nimotuzumab + SHR-1210

INTERVENTIONS:
Drug: Nimotuzumab + SHR-1210 — SHR-1210: 200 mg/time, intravenous injection, q2W continuous medication, a course of treatment needs 28 days. The cumulative longest medication period is 2 years.
  Nimotuzumab: 200 mg/time, intravenous injection, administered on the 1st and 8th days of each cycle, every 2 weeks is one cycle.

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of anti-PD-1 antibody SHR-1210 combined with nimotuzumab as second-line therapy in patients with advanced cancerous esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
The incidence of esophageal cancer is ranked seventh in the world, and the mortality rate ranks sixth in the world. At present, the first-line treatment of advanced esophageal cancer is mainly based on the combination of paclitaxel, cisplatin and fluorouracil. After the failure of first-line treatment, there is no standard second-line treatment. The investigators designed a single-arm, open phase II clinical trial of anti-PD-1 antibody SHR-1210 combined with nimotuzumab as second-line therapy in patients with advanced cancerous esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. 18~75 years, both men and women.
2. Pathologically (histologically or cytologically) confirmed diagnosis of esophageal squamous cell carcinoma (ESCC)， and locally advanced unresectable, local recurrence or distant metastasis.
3. Patients undergoing first-line systemic chemotherapy (which may include platinum, lavender or fluorouracil) progression or intolerance (progress in maintenance therapy after first-line chemotherapy can also be included). Synchronous chemoradiotherapy for postoperative recurrence or metastasis is considered as first-line treatment; For radical concurrent chemoradiotherapy, neoadjuvant/adjuvant therapy (chemotherapy or chemoradiotherapy), if disease progression occurs during treatment or within 6 months after stopping treatment, Count it as a first-line treatment failure.
4. At least one measurable/evaluable lesion by RECIST v1.1. And the measurable lesions should not have received local treatment such as radiotherapy (The lesion located in the previous radiotherapy area, if confirmed to progress, and meets the RECIST 1.1 standard, can also be used as a target lesion).
5. EGFR immunohistochemistry or FISH detection was positive in tumor tissue samples.
6. Tissue samples shall be provided for biomarker analysis, preferably newly acquired tissues, and patients who are unable to provide newly acquired tissues may provide 5-8 pieces of 5um thick paraffin sections that are archived and preserved.
7. Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1.
8. Life expectancy of ≥ 12 weeks.
9. The main organs function normally, that is, the following criteria are met:

(1) Blood routine examination:

1. HB≥90g/L;
2. ANC ≥ 1.5 × 109 / L;
3. PLT ≥ 80 × 109 / L. (2) Biochemical examination:

a. ALB ≥ 30g / L; b. ALT and AST ≤ 2.5ULN; if there is liver metastasis, ALT and AST ≤ 5ULN; c. TBIL ≤ 1.5ULN; d. plasma Cr ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min. 10. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF)≥ normal low limit (50%).

11. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months of the end of the study; the serum or urine pregnancy test is negative within 7 days prior to study enrollment, and Must be non-lactating; males should agree to use contraceptives during the study period and within 6 months of the end of the study period.

12. Subjects voluntarily joined the study, signed informed consent, and were well-adhered to follow-u.

Exclusion Criteria:

1. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroid Hyperfunction; patients with vitiligo; complete remission of asthma in childhood, can be included without any intervention after adult; asthma patients who require bronchodilators for medical intervention cannot be included).
2. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppression purposes (dose >10 mg/day of prednisone or other therapeutic hormones) and continues to be used within 2 weeks prior to enrollment.
3. Patients who received EGFR monoclonal antibody or EGFR tyrosine kinase inhibitor;
4. Patients who received other PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1;
5. Patients with brain metastases with symptoms or symptom control for less than 3 months;
6. Patients with any severe and/or uncontrolled diseases, including patients with unsatisfactory blood pressure control (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg); patients with grade I or higher myocardial ischemia or myocardial infarction, arrhythmia (including QT interval ≥ 480ms) and grade I cardiac insufficiency; active or uncontrolled severe infection; liver disease such as decompensated liver disease, active hepatitis B (HBV-DNA ≥ 104 copy number / ml or 2000 IU / ml) Or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the lower limit of detection of the analytical method);
7. Imaging studies have shown that the tumor has invaded the important vascular circumference or that the patient is likely to invade the important;
8. Pregnant or lactating women.
9. Patients with other malignant tumors within 5 years（Except for skin basal cell carcinoma and cervical carcinoma in situ that have been cured).
10. Patients with a history of psychotropic substance abuse who are unable to quit or have a mental disorder.
11. Patients who have participated in other drug clinical trials within four weeks.
12. According to the investigator's judgment, the patients with concomitant diseases that seriously endanger the safety of the patient or affect the patient's completion of the study.
13. Researchers believe that it is not suitable for inclusion. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 1 year
  From date of randomization until the date of death from any cause

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 1 year
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD)
Progression-free Survival (PFS) | up to 2 year
  From date of randomization until the date of first documented progression or date of death from any cause
Duration of response (DOR) | up to 2 year
  Refers to the time when the tumor is first evaluated as CR or PR until the first assessment is PD (Progressive Disease) or any cause of death.
Time to response (TTR) | up to 1 year
Overall survival(OS) | up to 2 year
  From date of randomization until the date of death from any cause
9-month survival rate | up to 9 month
12-month survival rate | up to 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Doctor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China